CLINICAL TRIAL: NCT02216227
Title: Checklist to Prevent MRSA Surgical Site Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRE 12-291
Record Dates: First submitted 2014-07-22; First posted 2014-08-13 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Surgical Site Infection
Keywords: MRSA; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Mupirocin; chlorhexidine gluconate; Chromogranins; Cefazolin; Vancomycin; Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Surgical Site Infection Checklist (Experimental): Patient has a known positive Staph aureus pre-op screening result (MRSA or MSSA):
  * ecolonize with intranasal Mupirocin ointment BID x 5 days
  * hlorhexidine gluconate (CHG) bathing (daily x 5 days, using wipes or liquid)
  * efazolin plus Vancomycin (no Vanco for MSSA positive)
  Patient has a known negative Staph aureus pre-op screening result:
  * HG bathing (night before & morning of surgery using wipes or liquid)
  * efazolin
  Patient was not screened or results are unknown at time of surgery:
  * ecolonize with intranasal Mupirocin ointment (start BID x 5 days; discontinue if negative screen)
  * HG bathing (start daily bath 5 days before operation if possible; at a minimum bathe the night before & morning of surgery using wipes or liquid)
  * efazolin plus Vancomycin
  Interventions: Drug: Mupirocin; Drug: Chlorhexidine gluconate; Drug: Cefazolin; Drug: Vancomycin; Drug: Nasal Povidone Iodine

INTERVENTIONS:
Drug: Mupirocin — Patients with known positive MRSA or MSSA and patients who have unknown status will decolonize BID x 5 days
  Other Names: Bactroban
Drug: Chlorhexidine gluconate — Patients that are MRSA or MSSA positive or have unknown status will bathe in CHG daily x 5 days.
  Patients that are MRSA or MSSA negative will bathe with CHG the night before and morning of surgery.
  Other Names: Chlorhexidine Gluconate in IMS, CHG
Drug: Cefazolin — All patients will receive Cefazolin during surgery
  Other Names: Ancef, Kefzol
Drug: Vancomycin — Patients who are positive for MRSA, or have unknown MRSA status, will receive vancomycin along with cefazolin during surgery.
  Other Names: vancocin
Drug: Nasal Povidone Iodine — The purpose of this research is to evaluate a SSI checklist. This checklist includes decolonizing a patient's nose and skin and optimizing antibiotics prior to surgery. At the time that we wrote it, the predominate product to decolonize patient's noses was mupirocin. However, in 2017, an FDA final monograph stated that nasal povidone-iodine may be used for pre-surgical decolonization. Nasal povidone-iodine should be able to overcome barriers to checklist implementation that we identified in Aim 3. We now plan to replace the nasal agent mupirocin with the nasal agent povidone-iodine at 3 participating medical centers (Iowa City VA, Minneapolis VA and Portland VA) to assess whether this overcomes the barriers to our SSI checklist.
  Other Names: Povidone Iodine

SUMMARY:
The goals of this project are 1) to assess the effectiveness and cost-effectiveness of the checklist to prevent MRSA SSIs among Veterans undergoing TJA or cardiac surgery, and 2) to assess barriers and facilitators to checklist implementation.

Hypotheses:

1. The SSI checklist will be effective at reducing MRSA SSIs among total joint arthroplasty and cardiac surgery patients.
2. Implementation of the checklist will be associated with an overall reduction in SSIs caused by all pathogens.
3. The SSI Checklist will be cost-saving since it will prevent many expensive SSIs.
4. Preoperative MRSA testing will be a modifiable barrier to implementing the SSI checklist.

DETAILED DESCRIPTION:
Aims and Design: Methicillin-resistant Staphylococcus aureus (MRSA), accounts for an estimated 94,000 invasive infections and 19,000 deaths annually in the U.S. In order to prevent MRSA infections among Veterans, the VA successfully implemented the VA MRSA Prevention Initiative that has reduced patient-to-patient transmission of MRSA. However, this Initiative does not prevent most MRSA surgical site infections (SSIs) because MRSA SSIs are usually caused by MRSA transferring from a patient's nose to their own surgical incision site. Cardiac surgery and total joint arthroplasty (TJA; e.g. hip or knee surgery) are among the most common operations performed by the VA and are associated with particularly high clinical and economic impact. In order to eliminate MRSA SSIs in the VA, the study group developed a checklist based on a meta-analysis of studies that assessed methods to prevent gram-positive SSIs among TJA and cardiac surgery patients. This SSI Checklist includes preoperatively testing a surgical patient's nose for asymptomatic MRSA colonization. If the patient is MRSA colonized, s/he will be treated with prophylactic nasal mupirocin ointment, chlorhexidine gluconate baths, and antibiotic prophylaxis with both cefazolin and vancomycin. The SSI Checklist will be implemented in 10 VA Medical Centers (VAMCs). A high-quality quasi-experimental study, with a qualitative process evaluation will be performed to assess the SSI Checklist. The goals of this project are 1) to assess the effectiveness and cost-effectiveness of the checklist to prevent MRSA SSIs among Veterans undergoing TJA or cardiac surgery, and 2) to assess barriers and facilitators to checklist implementation.

Methods: This study includes both quantitative and qualitative components. In the quantitative component, the SSI Checklist will be implemented in 10 VAMCs for 3 years and outcomes will be compared between the intervention group and two control groups: 1) 5 years of historic data from the same 10 VAMCs, 2) 8 years (5 historic year and 3 intervention years) of concurrent data from other VAMCs that did not implement the SSI Checklist. Study endpoints will include: 1) MRSA SSIs as defined by the Centers for Disease Control and Prevention (CDC); 2) SSIs caused by other pathogens; 3) cost per SSI prevented, cost per life-saved, cost per MRSA SSI prevented and cost per quality-adjusted life-year (QALY) saved. VA databases including VA National Surgical Quality Improvement Program (VASQIP), VA Decision Support System, VA Inpatient Evaluation Center (IPEC) and Veterans' Informatics & Computing Infrastructure (VINCI) will be used to collect data. Time series analysis and linear mixed effects models will be used for the statistical analysis. In the qualitative component, a process evaluation will be conducted at 6 different VAMCs, which includes collecting data before, during and after implementation, to examine the contextual factors and stakeholder perspectives that influence adoption of the SSI Checklist. Observations and semi-structured interviews will be conducted in Years 1 and 3, along with thematic content analysis, to examine facilitators and barriers to the implementation at the different study sites. The Consolidated Framework for Implementation Research will be used to guide the process evaluation and provide the foundation for a systematic evaluation of local contextual factors that influence implementation of the SSI Checklist. The products of this study include a validated SSI Checklist, a business-case analysis, an implementation toolkit, and a team experienced in checklist implementation for prevention of infections. At the end of this study period, the study team will meet with operational partners including National Infectious Disease Program Office (NIDS) and the MRSA / Multidrug-resistant Program Office (MDRO), and the National Center for Occupational Health and Infection Control (COHIC) to discuss implementing this checklist nationwide as part of the VA MRSA Prevention Initiative. This study has high potential to significantly decrease SSI, and in turn morbidity and mortality due to SSIs, in our Nation's Veterans.

ELIGIBILITY:
Inclusion Criteria:

Retrospective Control Group Inclusion Criteria:

* Patients identified in VA databases (e.g. VASQIP) by ICD-9 procedure codes as undergoing total joint arthroplasty or cardiac surgery at the 10 intervention VA Medical Centers during the 5 year preintervention period (2008-2013)

Concurrent Non-equivalent Control Group Inclusion Criteria:

* Patients identified in VA databases (e.g. VASQIP) by ICD-9 procedure codes as undergoing total joint arthroplasty or cardiac surgery at VA Medical Centers not included in the intervention group during the 8 years evaluated (5 years pre-intervention to match with the retrospective control group and 3 years of the intervention.)

Exclusion Criteria:

For All Patient Groups:

* Have an ICD-9 diagnosis code consistent with endocarditis
* Have any documented infection before the surgical procedure
* Undergo cardiac transplants or cardiac procedures performed using the percutaneous or thoracotomy approach
* Undergoing hip and knee revisions
* Documented allergies to mupirocin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1794 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Superficial and deep/organ space MRSA infections | 90 days postoperatively
  Superficial and deep/organ space MRSA infections, 90 days postoperatively.

SECONDARY OUTCOMES:
Superficial and deep/organ space MRSA infections | one year postoperatively
  The investigators chose 90-days rather than 1 year for the primary outcome measure since not all patients in the study will be able to be followed for 1 year due to the timing of the study. However, since the investigators will be able to follow 83% of the cohort for 1-year post-operatively, the investigators will perform this secondary analysis in which the investigators will include only patients who were followed for one year. However, it is unlikely that the 90-day analysis and 1 year analysis will differ significantly because over 75% of SSIs are detected within 30 days, in fact most SSI manifest within 22 days.
Compliance with the entire pre-surgical bundle and individual bundle components | 30-days pre-surgery to day of surgery
  This will be established electronically, through measurement of mupirocin prescription, CHG prescription and swab collection, as well as utilizing the compliance information collected on patient intake on the day of surgery.
Length of postoperative stay | Duration of postoperative stay, an expected average of 3 days
  Duration of postoperative stay, an expected average of 3 days.
All-cause mortality | Up to 1-year post-surgery
  All-cause mortality, Up to 1-year post-surgery.
Readmission | 90-days postsurgery
  Readmission, 90-days postsurgery.
Mupirocin and Chlorhexidine resistance in MRSA positive bacterial isolates | 30-days pre-surgery to 90-days post-surgery
  The investigators will test bacterial isolates from MRSA positive patients at the 10 interventions sites. The VA is mandated to take nasal swabs from each patient preoperatively. For those patients who are MRSA positive, the investigators will have the bacterial isolates sent to the Iowa City site to be tested for resistance to mupirocin and CHG. The investigators will also collect bacterial isolates from patients who experience surgical site infections during the study. These isolates will also be tested for mupirocin and CHG resistance.
  The purpose of this testing is to a) ensure the investigators' study checklist does not cause mupirocin or CHG resistance by b) determining if resistance was present at the initial nasal swab, or if resistance occurred after performance of study checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Eli N. Perencevich, MD MS BS, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (11):
- United States (11):
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrel M, Goto M, Schweizer ML, David MZ, Livorsi D, Perencevich EN. Diffusion of clindamycin-resistant and erythromycin-resistant methicillin-susceptible Staphylococcus aureus (MSSA), potential ST398, in United States Veterans Health Administration Hospitals, 2003-2014. Antimicrob Resist Infect Control. 2017 Jun 5;6:55. doi: 10.1186/s13756-017-0212-1. eCollection 2017. PMID 28593043
- [Background] Goto M, Schweizer ML, Vaughan-Sarrazin MS, Perencevich EN, Livorsi DJ, Diekema DJ, Richardson KK, Beck BF, Alexander B, Ohl ME. Association of Evidence-Based Care Processes With Mortality in Staphylococcus aureus Bacteremia at Veterans Health Administration Hospitals, 2003-2014. JAMA Intern Med. 2017 Oct 1;177(10):1489-1497. doi: 10.1001/jamainternmed.2017.3958. PMID 28873140
- [Background] Safdar N, Perencevich E. Crossing the quality chasm for Clostridium difficile infection prevention. BMJ Qual Saf. 2015 Jul;24(7):409-11. doi: 10.1136/bmjqs-2015-004344. Epub 2015 May 15. No abstract available. PMID 25979001
- [Result] Singh N, Nair R, Goto M, Carvour ML, Carnahan R, Field EH, Lenert P, Vaughan-Sarrazin M, Schweizer ML, Perencevich EN. Risk of Recurrent Staphylococcus aureus Prosthetic Joint Infection in Rheumatoid Arthritis Patients-A Nationwide Cohort Study. Open Forum Infect Dis. 2019 Oct 19;6(11):ofz451. doi: 10.1093/ofid/ofz451. eCollection 2019 Nov. PMID 31737738
- [Result] Pfeiffer CD, Williams HB, Flegal H, Klutts JS, Evans M, Jones MM. 493. Laboratory Evaluation and Epidemiology of Carbapenemase-Producing Carbapenem-Resistant Enterobacteriaceae in Department of Veterans Affairs, 2017. [Abstract]. Open forum infectious diseases. 2019 Oct 23; 6(Supplement_2):S240-S241.
- [Derived] Hockett Sherlock S, Goedken CC, Balkenende EC, Dukes KC, Perencevich EN, Reisinger HS, Forrest GN, Pfeiffer CD, West KA, Schweizer M. Strategies for the implementation of a nasal decolonization intervention to prevent surgical site infections within the Veterans Health Administration. Front Health Serv. 2022 Aug 17;2:920830. doi: 10.3389/frhs.2022.920830. eCollection 2022. PMID 36925849